CLINICAL TRIAL: NCT05978505
Title: Reboxetine for Obstructive Sleep Apnoea After Upper Airway Surgery: a Randomised, Double-blind, Placebo-controlled Study
Brief Title: Reboxetine for Sleep Apnoea After ENT Surgery
Acronym: RENTOSA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Flinders University (Other)
Collaborators: Flinders Medical Centre (Other Government)
Responsible Party: Principal Investigator, Professor Danny Eckert, Director, Adelaide Institute for Sleep Health, Flinders University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 2023/HRE00060
Record Dates: First submitted 2023-06-02; First posted 2023-08-07 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Sleep Apnea, Obstructive
Keywords: sleep apnea, obstructive; upper airway surgery; ENT surgery; reboxetine; noradrenaline reuptake inhibitor; randomised; feasibility; placebo; double-blind
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Reboxetine; Tablets; Sugars

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo-controlled, cross-over study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Identical capsule for placebo and study drug prepared by study pharmacist
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Reboxetine (Experimental): 7-day course of 4mg reboxetine, taken nightly before bed time. Reboxetine will be taken for 7-nights post-surgery.
  Interventions: Drug: Reboxetine 4 MG Oral Tablet
- Placebo (Placebo Comparator): Placebo sugar pill in the form of one capsule, taken before bedtime. Dosage is taken for 7 nights post-surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Reboxetine 4 MG Oral Tablet — 7 nightly doses (4mg) to commence after surgery.
  Other Names: Edronax
  Arms: Reboxetine
Drug: Placebo — 7 nightly doses to commence after surgery.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
This pilot study will establish the feasibility of a larger trial to investigate whether reboxetine, a medication used to treat depression, can reduce the severity of obstructive sleep apnea (OSA) including increased blood oxygenation in post-surgical OSA patients where positive airway pressure (CPAP) therapy is either frequently poorly tolerated or not an option immediately post surgery. In this randomized, placebo-controlled, double-blind study, participants will use at-home sleep monitoring equipment before and after surgery plus measures of oxygenation. They will be prescribed either reboxetine or a placebo for seven days after surgery and complete questionnaires at the beginning and end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Undergoing elective upper airway surgery
* History of obstructive sleep apnoea (OSA)

Exclusion Criteria:

* Clinically significant cardiac disease (e.g., arrhythmia, coronary artery disease, or cardiac failure)
* History of clinically significant urinary retention, bladder outlet obstruction, or benign prostatic hyperplasia
* Poorly controlled hypertension
* Epilepsy
* History of schizophrenia, schizoaffective disorder or bipolar disorder according to Diagnostic and Statistical Manual of Mental Disorders-V or International Classification of Disease 10th edition criteria
* History of attempted suicide or suicidal ideation within 1 year prior to screening, or current suicidal ideation
* Narrow angle glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Treatment protocol adherence | 7 days
  The percentage of total doses of the study drug (reboxetine or placebo) that were taken versus prescribed (assessed via pill counts) for this feasibility study.
Data capture efficiency | 14 days
  The percentage of successful data collection nights versus missed nights of at-home oximetry for this feasibility study.

SECONDARY OUTCOMES:
Oxygen desaturation index (ODI) | 14 days
  Number of times per hour that a participant has a drop in blood oxygen levels during sleep
nadir SpO2 | 14 days
  The lowest oxygen saturation value the patient drops to in a night.
Time spent below 90% SpO2 | 14 days
  The total amount of time per night for which oxygen saturation falls below 90%.
mean SpO2 | 14 days
  Average nightly oxygen level
Sleep duration | 14 days
  Total amount of time spent asleep per night, sleep tracking performed using an under mattress sensor device.
Sleep efficiency (%) | 14 days
  The estimated percentage of time in bed spent asleep performed using an under mattress sensor device.
Daytime sleepiness | 14 days
  Measured via Karolinska Sleepiness Scale Questionnaire (9 point scale where 1 = extremely alert and 9 = extremely sleepy - fighting sleep)
Perceived sleep quality measured via the Leeds Sleep Evaluation Questionnaire | 14 days
  This questionnaire asks participants to rate their perceived sleep across 4 domains on a visual analog scale as follows: 1) getting to sleep, 2) quality of sleep, 3) Awake following sleep, 4) Behavior following wakening. Higher scores indicate better perceived sleep.
Insomnia Severity Score | 14 days
  A patient-reported measure of insomnia symptoms using the Insomnia Severity Index- A 28 point scale where 0 indicates no clinically significant insomnia and 28 indicates maximally severe clinical insomnia.
Apnoea-hypopnea hndex (AHI) | 14 days
  Change in OSA severity (AHI estimated via the Withings under mattress sensor number of events/hour) between placebo and reboxetine
Study enrolment rate | 12 months
  The number of referred patients successfully enrolled into this feasibility study

OTHER OUTCOMES:
Reboxetine-related side effects | 14 days
  Documented via adverse-event forms.

CONTACTS AND LOCATIONS:
Overall Officials: Danny J. Eckert, PhD, Principal Investigator — Flinders University
Locations (1):
- Flinders, Private and Public Hospitals and Flinders University, Bedford Park, South Australia, Australia

IPD SHARING:
Plan to Share IPD: Yes
Participants will be informed in plain language through the consent form that their deidentified data may be made available to other researchers. Deidentified participant data will only be shared with other researchers upon request to the chief investigator after study publication and subject to ethical approval
Supporting Information: Study Protocol, ICF
Time Frame: At conclusion of the study and any related publications
Access Criteria: IPD may be shared for research purposes on application to the chief investigator and subject to applicable ethical review.

REFERENCES:
- [Background] Opperer M, Cozowicz C, Bugada D, Mokhlesi B, Kaw R, Auckley D, Chung F, Memtsoudis SG. Does Obstructive Sleep Apnea Influence Perioperative Outcome? A Qualitative Systematic Review for the Society of Anesthesia and Sleep Medicine Task Force on Preoperative Preparation of Patients with Sleep-Disordered Breathing. Anesth Analg. 2016 May;122(5):1321-34. doi: 10.1213/ANE.0000000000001178. PMID 27101493
- [Background] Chan MTV, Wang CY, Seet E, Tam S, Lai HY, Chew EFF, Wu WKK, Cheng BCP, Lam CKM, Short TG, Hui DSC, Chung F; Postoperative Vascular Complications in Unrecognized Obstructive Sleep Apnea (POSA) Study Investigators. Association of Unrecognized Obstructive Sleep Apnea With Postoperative Cardiovascular Events in Patients Undergoing Major Noncardiac Surgery. JAMA. 2019 May 14;321(18):1788-1798. doi: 10.1001/jama.2019.4783. PMID 31087023
- [Background] Khanna AK, Bergese SD, Jungquist CR, Morimatsu H, Uezono S, Lee S, Ti LK, Urman RD, McIntyre R Jr, Tornero C, Dahan A, Saager L, Weingarten TN, Wittmann M, Auckley D, Brazzi L, Le Guen M, Soto R, Schramm F, Ayad S, Kaw R, Di Stefano P, Sessler DI, Uribe A, Moll V, Dempsey SJ, Buhre W, Overdyk FJ; PRediction of Opioid-induced respiratory Depression In patients monitored by capnoGraphY (PRODIGY) Group Collaborators. Prediction of Opioid-Induced Respiratory Depression on Inpatient Wards Using Continuous Capnography and Oximetry: An International Prospective, Observational Trial. Anesth Analg. 2020 Oct;131(4):1012-1024. doi: 10.1213/ANE.0000000000004788. PMID 32925318
- [Background] Altree TJ, Eckert DJ. Obstructive sleep apnea endotypes and their postoperative relevance. Int Anesthesiol Clin. 2022 Apr 1;60(2):1-7. doi: 10.1097/AIA.0000000000000357. No abstract available. PMID 35125480
- [Background] Chung F, Liao P, Yegneswaran B, Shapiro CM, Kang W. Postoperative changes in sleep-disordered breathing and sleep architecture in patients with obstructive sleep apnea. Anesthesiology. 2014 Feb;120(2):287-98. doi: 10.1097/ALN.0000000000000040. PMID 24158049
- [Background] Chung F, Memtsoudis SG, Ramachandran SK, Nagappa M, Opperer M, Cozowicz C, Patrawala S, Lam D, Kumar A, Joshi GP, Fleetham J, Ayas N, Collop N, Doufas AG, Eikermann M, Englesakis M, Gali B, Gay P, Hernandez AV, Kaw R, Kezirian EJ, Malhotra A, Mokhlesi B, Parthasarathy S, Stierer T, Wappler F, Hillman DR, Auckley D. Society of Anesthesia and Sleep Medicine Guidelines on Preoperative Screening and Assessment of Adult Patients With Obstructive Sleep Apnea. Anesth Analg. 2016 Aug;123(2):452-73. doi: 10.1213/ANE.0000000000001416. PMID 27442772
- [Background] Liao P, Luo Q, Elsaid H, Kang W, Shapiro CM, Chung F. Perioperative auto-titrated continuous positive airway pressure treatment in surgical patients with obstructive sleep apnea: a randomized controlled trial. Anesthesiology. 2013 Oct;119(4):837-47. doi: 10.1097/ALN.0b013e318297d89a. PMID 24195872
- [Background] Altree TJ, Chung F, Chan MTV, Eckert DJ. Vulnerability to Postoperative Complications in Obstructive Sleep Apnea: Importance of Phenotypes. Anesth Analg. 2021 May 1;132(5):1328-1337. doi: 10.1213/ANE.0000000000005390. PMID 33857975
- [Background] Reilly EK, Boon MS, Vimawala S, Chitguppi C, Patel J, Murphy K, Doghramji K, Nyquist GG, Rosen MR, Rabinowitz MR, Huntley CT. Tolerance of Continuous Positive Airway Pressure After Sinonasal Surgery. Laryngoscope. 2021 Mar;131(3):E1013-E1018. doi: 10.1002/lary.28968. Epub 2020 Sep 16. PMID 32936959
- [Background] Perger E, Taranto Montemurro L, Rosa D, Vicini S, Marconi M, Zanotti L, Meriggi P, Azarbarzin A, Sands SA, Wellman A, Lombardi C, Parati G. Reboxetine Plus Oxybutynin for OSA Treatment: A 1-Week, Randomized, Placebo-Controlled, Double-Blind Crossover Trial. Chest. 2022 Jan;161(1):237-247. doi: 10.1016/j.chest.2021.08.080. Epub 2021 Sep 20. PMID 34543665
- [Background] Taranto-Montemurro L, Messineo L, Sands SA, Azarbarzin A, Marques M, Edwards BA, Eckert DJ, White DP, Wellman A. The Combination of Atomoxetine and Oxybutynin Greatly Reduces Obstructive Sleep Apnea Severity. A Randomized, Placebo-controlled, Double-Blind Crossover Trial. Am J Respir Crit Care Med. 2019 May 15;199(10):1267-1276. doi: 10.1164/rccm.201808-1493OC. PMID 30395486
- [Background] Lim R, Messineo L, Grunstein RR, Carberry JC, Eckert DJ. The noradrenergic agent reboxetine plus the antimuscarinic hyoscine butylbromide reduces sleep apnoea severity: a double-blind, placebo-controlled, randomised crossover trial. J Physiol. 2021 Sep;599(17):4183-4195. doi: 10.1113/JP281912. Epub 2021 Jul 14. PMID 34174090